CLINICAL TRIAL: NCT00764933
Title: A Randomized Controlled Multi Center Study to Evaluate the Efficacy of a Structured Information Program During ICU Stay
Brief Title: Structured Information During the Intensive Care Unit Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. phil habil Johann Behrens, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PfVMS-T4
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-01

CONDITIONS: Anxiety
Keywords: information programme; anxiety reduction; multicenter trial; intensive care; critical care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Structured information
  Interventions: Behavioral: Structured information
- 2 (Sham Comparator): Unspecific conversation
  Interventions: Other: Unspecific conversation

INTERVENTIONS:
Behavioral: Structured information — Participants will receive structured information about their ICU-stay and course of therapy and care. They get information about procedures, sensory impressions and coping strategies. The intervention will last about 10 to 15 minutes depending on the state of the participant.
  Arms: 1
Other: Unspecific conversation — Participants will receive a short conversation with the study personnel. This conversation will last about 10 to 15 minutes. No specific informations will be given about procedures, sensory impressions or coping strategies. Control intervention is designed to control for personal attention and care.
  Arms: 2

SUMMARY:
The purpose of this study is to test whether a structured information program at the beginning of the ICU-stay is effective to reduce ICU related anxiety and discomfort.

DETAILED DESCRIPTION:
The trial is designed as a prospective multicenter randomized controlled trial including an intervention and a control group. The control group receives an unspecific conversation. The intervention group receives a standardized information program with specific procedural, sensory and coping information about the ICU. Anxiety will be measured with a VAS during ICU stay and with a questionnaire after ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Elective open heart or abdominal surgery including scheduled ICU stay
* Heart or abdominal surgery or internal patients with non-scheduled ICU stay
* Informed consent

Exclusion Criteria:

* Reduced sensual perception
* Cognitive impairment
* Not able to answer a questionnaire (e.g. illiterate)
* Lying in the same room with another patient already included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Patient self-reported anxiety | First three days on ICU and/or within 24 hours after ICU discharge

SECONDARY OUTCOMES:
Confusion Assessment Method for the ICU (CAM-ICU) | Within first three days on ICU
Patient self reported health-related quality of life | 3 months after discharge from hospital

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Sana Herzchirurgische Klinik Stuttgart GmbH, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Gießen und Marburg, Kooperationsstudien Pflegedienst/Ärztlicher Dienst, Klinik für Visceral-, Thorax- und Gefäßchirurgie, Klinik für Herz- und thorakale Gefäßchirurgie, Standort Marburg, Marburg, Hesse
  - Institut für Gesundheits- und Pflegewissenschaft, Universitätsklinik für Anästhesiologie und operative Intensivmedizin, Medizinische Fakultät, Martin-Luther-Universität Halle-Wittenberg, Halle, SAN

REFERENCES:
- [Derived] Fleischer S, Berg A, Behrens J, Kuss O, Becker R, Horbach A, Neubert TR. Does an additional structured information program during the intensive care unit stay reduce anxiety in ICU patients?: a multicenter randomized controlled trial. BMC Anesthesiol. 2014 Jun 28;14:48. doi: 10.1186/1471-2253-14-48. eCollection 2014. PMID 25071414
- [Derived] Fleischer S, Berg A, Neubert TR, Koller M, Behrens J, Becker R, Horbach A, Radke J, Rothmund M, Kuss O. Structured information during the ICU stay to reduce anxiety: study protocol of a multicenter randomized controlled trial. Trials. 2009 Sep 14;10:84. doi: 10.1186/1745-6215-10-84. PMID 19751500